CLINICAL TRIAL: NCT00684424
Title: Non-Interventional Study (NIS) With Lyrica In Patients With Epilepsy As Adjunctive Therapy Of Partial Seizures To Reduce Seizure Frequency
Brief Title: Non-Interventional Study With LYRICA (Pregabalin) In Patients With Epilepsy As Adjunctive Therapy Of Partial Seizures To Reduce Seizure Frequency
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081213
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2010-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients with epilepsy
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Observational Only

SUMMARY:
The primary efficacy parameter will be the responder rate, defined as the proportion of subjects who had at least a 50% reduction in 28 day seizure rate during the maintenance phase

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old, patients with epilepsia with partial seizures
* Enrollment to study is fully on physician decision in compliance with current SPC.

Exclusion Criteria:

* Patient who did not meet indication according to SPC Lyrica

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081213&StudyName=Non-Interventional%20Study%20with%20LYRICA%AE%20In%20Patients%20With%20Epilepsy%20As%20Adjunctive%20Therapy%20Of%20Partial%20Seizures%20To%20Reduce%20Seizure%20Frequency%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 36 medical centers and participated in the study between 11 July 2008 and 30 March 2009.
Groups:
- Pregabalin (Lyrica): Individualized dose ranging from 150 mg to 600 mg daily administered as two single doses.
Period: Overall Study
Arm/Group | Pregabalin (Lyrica)
Started | 199
Completed | 194
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
Age, Customized [Number; unit: participants]
  <=18 years | 2
  18 - 44 years | 104
  45 - 65 years | 60
  >= 65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 92

OUTCOME MEASURES:

1. Primary Outcome: Responders: Number of Subjects With a 50% or Greater Reduction in Seizure Frequency
Description: Responders: number of subjects with a 50 percent (%) or greater reduction in partial seizure frequency from Baseline to Final visit. Seizure frequency in treatment period = total number of partial seizures in maintenance treatment phase * 28 divided by total number of days in the maintenance treatment phase. Missing category includes subjects with missing attack date, insufficient length of treatment period or no seizures in both baseline and treatment periods. Subjects with zero seizures in the baseline period and some seizures in the treatment period were treated as non-responders.
Time Frame: Baseline through Week 16
Population: Full Analysis Set: all subjects who received at least 1 dose of study drug and had at least 1 efficacy measurement.
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Responders | 138
  Non-Responders | 44
  Missing | 17

2. Secondary Outcome: Antiepileptic Drugs Used in the Past
Description: Antiepileptic drug history: number of subjects who took each class of antiepileptic drug prior to entering the study. Subjects who took more than one antiepileptic drug were counted for each of the drug classes.
Time Frame: Baseline
Population: Safety analysis set: all subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Barbiturates | 42
  Carbamazepine | 93
  Gabapentin | 30
  Lamotrigine | 38
  Levetiracetam | 26
  Phenytoin | 66
  Tiagabine | 4
  Topiramate | 40
  Valproate | 97
  Vigabatrine | 4
  Other | 16
  Missing | 9
  No previous treatment | 11

3. Secondary Outcome: Change in 28 Day Partial Seizure Frequency
Description: Change in 28-day partial seizure frequency between the baseline period and treatment period. Baseline period = the 4 weeks (28 days) prior to Baseline visit. Treatment period = last 12 weeks (84 days) of the study (maintenance treatment phase excluding 4-week titration phase). Seizure frequency in baseline period = total number of partial seizures in baseline phase * 28 divided by total number of days in the baseline phase. Seizure frequency in treatment period = total number of partial seizures in maintenance treatment phase * 28 divided by total number of days in maintenance treatment phase.
Time Frame: Baseline through Week 16 (Final Visit )
Population: FAS. Subjects who discontinued less than 4 weeks into the treatment period or with missing date of the attack were excluded from analyses.
Measure: Mean (Standard Deviation); unit: number of seizures per 28 days
Arm/Group | Pregabalin
Number analyzed (Participants) | 196
number of seizures per 28 days
  Baseline Period | 3.20 (3.375)
  Treatment Period | 1.339 (2.5177)
  Change from Baseline to Treatment Period | -1.860 (2.0494)
Statistical Analysis 1: Comparison: Pregabalin; R-ratio of seizure frequency summaries = [(t-b)/(t+b)]*100; where t= treatment seizure frequency and b= baseline seizure frequency; Test type: Superiority or Other; summary statistic; R-ratio = -56.723, Standard Deviation 46.9499

4. Secondary Outcome: Seizure Freedom: Number of Seizure-free Subjects During the Last 4 Weeks of the Study
Description: Seizure Freedom (responders): subjects with no seizures (partial or other) during the last 4 weeks of the study. Non-responders: subjects with seizures (partial or other)during the last 4 weeks of the study. Subjects, who discontinued less than 4 weeks into the observation period were excluded from analysis. The 4 week period excludes the titration phase of the study. Missing category includes subjects with missing attack date or insufficient length of treatment period.
Time Frame: Week 8 up to Week 16 (Last 4 weeks of the treatment period)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Responders: Seizure-free | 119
  Non-responders: With Seizures | 77
  Missing | 3

5. Secondary Outcome: Concomitant Drug Treatments
Description: Concomitant drugs treatments (drugs other than, and in addition to study medication): number of subjects who took each concomitant drug during the study (baseline through end of study). World Health Organization (WHO) Drug (v02Q2) coding dictionary applied.
Time Frame: Baseline through Week 16 (Final Visit)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Acetylsalicylic acid | 2
  Acidum folicum | 1
  Alendronic acid | 1
  Alprazolam | 2
  Amlodipine besilate | 1
  Amlozek | 1
  Anopyrin | 3
  Atorvastatin calcium | 1
  Aurorix | 1
  Biston | 1
  Carbamazepine | 26
  Cipralex | 1
  Citalopram | 2
  Citalopram hydrobromide | 1
  Clonazepam | 6
  Colecalciferol | 1
  Depakine | 10
  Depakine chrono | 14
  Detralex | 1
  Diarel | 1
  Diazepam | 1
  Dipyridamole | 1
  Enelbin - slow release | 1
  Euthyrox | 2
  Felodipine/ramipril | 1
  Fenytoin | 1
  Fluanxol depot | 1
  Gabapentin | 3
  Gabitril | 1
  Geratam | 1
  Ginko biloba | 1
  Glibenclamide | 1
  Glucobene | 1
  Godasal | 2
  Hypnogen | 1
  Keppra | 20
  Lamictal | 18
  Lamotrigine | 49
  Letrox | 2
  Levetiracetam | 20
  Levothyroxine | 2
  Lexaurin | 1
  Lipanthyl | 2
  Lispril | 1
  Liskantin | 4
  Lokren | 1
  Lusopress | 1
  Magnesium | 1
  Magnesium lactate | 2
  Metformin | 1
  Metoprolol | 1
  Micardis | 2
  Neurontin | 1
  Neurotop | 3
  Neurotop - slow release | 5
  Omeprazol | 1
  Omeprazole | 1
  Paroxetine | 1
  Pentomer | 1
  Perindopril | 1
  Perindopril erbumine | 1
  Phenytoin | 4
  Piracetam | 2
  Prestarium | 5
  Primdone | 2
  Ramipril | 1
  Ramipril/hydrochlorothiazide | 1
  Rivotril | 8
  Rufinamide | 1
  Sabril | 1
  Sanepil | 1
  Seretide diskus | 1
  Sertraline | 1
  Simepar | 1
  Simvastatin | 1
  Siofor | 1
  Sodanton | 1
  Sorbimon | 1
  Sumatriptan | 1
  Symbicort turbuhaler "Draco" | 1
  Tegretol | 2
  Tegretol CR | 8
  Ticlopidine | 3
  Timonil | 1
  Timonil - slow release | 8
  Topamax | 15
  Topiramate | 25
  Trandlapril | 1
  Valproate | 22
  Valproate sodium | 7
  Valproic acid | 14
  Vasocardin | 1
  Vinpocetine | 1
  Warfarin | 1
  Zocor | 2
  Zoloft | 1

6. Secondary Outcome: Average Dosage of Pregabalin Taken at Baseline and Final Visit
Description: Average doses of pregabalin in milligrams per day (mg/day) taken at baseline and final visit shown by number of participants at each dose.
Time Frame: Baseline, Week 16 (Final Visit )
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Baseline: 75 mg | 31
  Baseline:100 mg | 0
  Baseline: 130 mg | 1
  Baseline: 150 mg | 166
  Baseline: 225 mg | 0
  Baseline: 300 mg | 1
  Baseline: 375 mg | 0
  Baseline: 450 mg | 0
  Baseline: 525 mg | 0
  Baseline: 600 mg | 0
  Final Visit: 75 mg | 8
  Final Visit: 100 mg | 1
  Final Visit: 130 mg | 1
  Final Visit: 150 mg | 55
  Final Visit: 225 mg | 5
  Final Visit: 300 mg | 89
  Final Visit: 375 mg | 1
  Final Visit: 450 mg | 6
  Final Visit: 525 mg | 1
  Final Visit: 600 mg | 32

7. Secondary Outcome: Visual Analog Scale of Anxiety (VAS-A)
Description: Visual Analog Scale of anxiety self assessment: metric measurement (in 2 mm interval) from the visual analog scale; 0 mm = no anxiety, 100 mm = extreme anxiety at each visit.
Time Frame: Baseline, Week 4, Week 16 (Final Visit), Last Observation Carried Forward
Population: FAS; Last observation carried forward (LOCF) method: subject's last available post-baseline observation was used if data were missing. In this case, data from Visit 2 were carried forward if final visit data were missing.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
mm
  Baseline (n=197) | 47.1 (21.52)
  Week 4 (Visit 2 ) (n=196) | 36.7 (18.43)
  Week 16 (Final Visit ) (n=197) | 29.0 (17.05)
  Last Observation Carried Forward (LOCF) (n=198) | 29.0 (17.03)

8. Secondary Outcome: Change From Baseline to Final Visit in Visual Analog Scale of Anxiety (VAS-A)
Description: Visual Analog Scale of anxiety self assessment: metric measurement (in 2 mm interval) from the visual analog scale; 0 mm = no anxiety, 100 mm = extreme anxiety. Change from Baseline to Final Visit: score at final visit minus score at baseline.
Time Frame: Baseline, Week 16 (Final Visit), Last Observation Carried Forward
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
mm
  Change from Baseline to Week 16 (n=196) | -18.2 (17.61)
  Change from Baseline to LOCF (n=197) | -18.1 (17.64)

9. Secondary Outcome: Number of Subjects With Categorical Scores on Clinical Global Impression of Severity (CGI-S)
Description: CGI-S scale: physician's global impression of a subject's clinical condition, at baseline in terms of severity. Numerical scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill subjects). Numbers of subjects in each category are presented.
Time Frame: Baseline
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Normal, not at all ill | 28
  Borderline mentally ill | 77
  Mildly ill | 39
  Moderately ill | 31
  Markedly ill | 14
  Severely ill | 9
  Among the most extremely ill patients | 1

10. Secondary Outcome: Number of Subjects With Categorical Scores on Clinical Global Impression of Change(CGI-C)
Description: CGI-C scale: physician's global impression of a subject's clinical condition in terms of change from baseline. Improvement = CGI response of very much improved, much improved, or minimally improved. No Change = CGI response of no change. Worsening = CGI response of very much worse, much worse or minimally worse.
Time Frame: Week 16 (Final Visit)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  Improvement | 174
  No Change | 21
  Worsening | 2
  Missing | 2

11. Secondary Outcome: Medical Outcomes Sleep Scale (MOS-S)
Description: MOS-S: subject reported measure with 12 items that assess key constructs of sleep over the past week. Scoring based on 7 subscales: sleep disturbance, snoring, awakened short of breath or with headache, sleep adequacy, and somnolence (range:0-100); sleep quantity (range:0-24), and optimal sleep (yes:1, no:0). Six(6) and 9 item index measures of sleep disturbance were constructed to provide composite scores. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range * 100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 16 (Final Visit )
Population: FAS. A subscale was classified as missing if any of the questions used in the calculation were missing. Abbreviations: BL = Baseline, SOB = short of breath.
Measure: Mean (Standard Deviation); unit: scores on scales
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
scores on scales
  Baseline: Sleep Disturbance | 37.86 (20.643)
  Baseline: Snoring | 29.1 (21.31)
  Baseline: Awaken Short of Breath or With Headache | 18.5 (19.26)
  Baseline: Quantity of Sleep | 7.0 (1.40)
  Baseline: Sleep Adequacy | 47.51 (24.336)
  Baseline: Somnolence | 35.99 (16.197)
  Baseline: Sleep 6-Item Index | 38.74 (17.522)
  Baseline: Sleep 9-Item Index | 38.82 (16.840)
  Final Visit: Sleep Disturbance | 25.21 (15.670)
  Final Visit: Snoring | 26.5 (21.86)
  Final Vst: Awaken Short of Breath or With Headache | 15.1 (16.68)
  Final Visit: Quantity of Sleep | 7.5 (1.31)
  Final Visit: Sleep Adequacy | 60.00 (22.113)
  Final Visit: Somnolence | 30.09 (15.398)
  Final Visit: Sleep 6-Item Index | 29.30 (14.501)
  Final Visit: Sleep 9-Item Index | 28.69 (13.399)
  Change from BL: Sleep Disturbance | -13.07 (17.010)
  Change from BL: Snoring | -2.9 (13.01)
  Change from BL: Awaken SOB or Headache | -3.8 (13.55)
  Change from BL: Quantity of Sleep | 0.6 (1.23)
  Change from BL: Sleep Adequacy | 13.02 (19.636)
  Change from BL: Somnolence | -6.18 (14.399)
  Change from BL: Sleep 6-Item Index | -9.88 (13.641)
  Change from BL: Sleep 9-Item Index | -10.54 (13.280)

12. Secondary Outcome: Number of Subjects With Change in Response Categories in Medical Outcomes Sleep Scale (MOS-S): Optimal Sleep Subscale
Description: MOS: subject rated questionnaire to assess sleep quality and quantity. Optimal sleep subscale is derived from Sleep Quantity average hours of sleep each night during the past week. Number of subjects with response: YES (Optimal) if sleep quantity was 7 or 8 hours per night, or response = NO (Non-Optimal) if sleep quantity was less than (<) 7 hours per night. Number of participants with shift in response categories from Baseline to Final Visit.
Time Frame: Baseline, Week 16 (Final Visit)
Population: FAS. Abbreviations: BL = Baseline; FV = Final Visit.
Measure: Number; unit: participants
Arm/Group | Pregabalin (Lyrica)
Number analyzed (Participants) | 199
participants
  BL: Optimal Sleep; FV: Optimal Sleep | 82
  BL: Optimal Sleep; FV: Non-Optimal Sleep | 10
  BL: Optimal Sleep; FV: Missing | 2
  BL: Non-Optimal Sleep; FV: Optimal Sleep | 33
  BL: Non-Optimal Sleep; FV: Non-Optimal Sleep | 48
  BL: Non-Optimal Sleep; FV: Missing | 5
  BL: Missing; FV: Optimal Sleep | 1
  BL: Missing; FV: Non-Optimal Sleep | 2
  BL: Missing; FV: Missing | 16

ADVERSE EVENTS:
Arm/Group | Pregabalin (Lyrica)
Serious Adverse Events (participants affected / at risk) | 1/199
Other Adverse Events (participants affected / at risk) | 26/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (Lyrica) (N=199)
Hemiplegia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (Lyrica) (N=199)
Vertigo (Ear and labyrinth disorders) | 2
Oedema peripheral (General disorders) | 1
Weight increased (Investigations) | 6
Dizziness (Nervous system disorders) | 10
Epilepsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.